CLINICAL TRIAL: NCT04488406
Title: Genetics and Epigenetics of Graves' Orbitopathy
Acronym: GeneGO
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Associate Professor, University of Pisa
Other Study IDs: GeneGO
Record Dates: First submitted 2020-07-17; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Graves' Orbitopathy: Graves' Orbitopathy patients who undergoing orbital decompressive surgery
  Interventions: Other: No Intervention
- Control Patients: Patients undergoing eye surgery for unrelated reasons
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Not applicable to these subjects. There is no study-related intervention

SUMMARY:
Graves' orbitopathy (GO) is an autoimmune disease persisting when immunosuppression is achieved. Orbital fibroblasts from GO patients display peculiar phenotypes even if not exposed to autoimmunity, possibly reflecting genetic or epigenetic mechanisms, to be investigated here.

Primary cultures of orbital fibroblasts from GO and control patients will be established. Cell proliferation, release of hyaluronic acid (HA) and HA synthases (HAS) will be measured. Next Generation Sequencing and gene expression analysis of the whole genome will be performed, as well as global DNA methylation assay.

DETAILED DESCRIPTION:
The investigators will establish primary cultures of orbital fibroblasts from orbital adipose tissue samples taken from six GO patients who underwent orbital decompressive surgery. Normal orbital tissue samples will be collected from six patients undergoing eye surgery for unrelated reasons.

Cell proliferation and HA will be measured using commercial assays DNA and RNA will be extracted. HAS-1, HAS-2 and HAS-3 will be measured were assessed by Real Time-PCR Next Generation Sequencing, Gene expression analysis and DNA methylation assays will be performed

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Graves' Orbitopathy
* Informed consent

Exclusion Criteria:

-Lack of informed consent

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Graves' orbitopathy undergoing decompressione surgery
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Gene expression | Baseline
  Gene expression in patients vs controls

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cisanello-Endocrinology I and II, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rotondo Dottore G, Bucci I, Lanzolla G, Dallan I, Sframeli A, Torregrossa L, Casini G, Basolo F, Figus M, Nardi M, Marcocci C, Marino M. Genetic Profiling of Orbital Fibroblasts from Patients with Graves' Orbitopathy. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2176-e2190. doi: 10.1210/clinem/dgab035. PMID 33484567